CLINICAL TRIAL: NCT06889038
Title: Hyperbaric Oxygen Therapy Combined With Polarized Light Therapy Effect on Neuropathic Foot Ulcer Regarding Transcutaneous Oxygen Saturation (TcpO2) and Healing Rate ( A Randomized Control Study)
Brief Title: Hyperbaric Oxygen Therapy Combined With Polarized Light Therapy Effect on Neuropathic Foot Ulcer
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Al-Zaytoonah University of Jordan (Other)
Responsible Party: Principal Investigator, Hanan Hosny M Battesha, associate professor, Al-Zaytoonah University of Jordan
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Hyperbaric oxygen therapy
Record Dates: First submitted 2025-03-15; First posted 2025-03-21 (Actual); Last update posted 2025-08-22 (Actual); Status verified 2025-08

CONDITIONS: Neuropathic Diabetic Ulcer - Foot
Keywords: Hyperbaric oxygen therapy; polarized light therapy; neuropathic foot ulcer

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- study group (Experimental): patients will evaluated to be fit for HBO therapy to ensure cardiac ejection fraction over 50% and chest CT to ensure chest free from any pathology
  Interventions: Other: Hyperbaric oxygen therapy combined with polarized light therapy
- control (Active Comparator): topical medication
  Interventions: Other: traditional treatment

INTERVENTIONS:
Other: Hyperbaric oxygen therapy combined with polarized light therapy — Optimum regime of therapy increase healing rate of neuropathic foot ulcer is a challenge for researchers to save patient normal life
  Arms: study group
Other: traditional treatment — topical medication
  Arms: control

SUMMARY:
Neuropathic ulcers develop due to nerve damage (neuropathy), commonly seen in conditions like diabetes, leading to loss of sensation, repetitive trauma, and poor wound healing. These ulcers typically occur on weight-bearing areas, hyperbaric oxygen and polarized light therapies may have a synergistic effect, improving oxygenation, cellular activity, and overall healing outcomes in neuropathic ulcers, particularly in diabetic foot ulcers.

ELIGIBILITY:
Inclusion Criteria:

* All patients had cardiac ejection fraction (CEF) 50%
* blood pressure (BP) 150/90mmHg.
* Chest X-ray was reported normal
* all patients were clinically evaluated by a specialized ear, nose, and throat (ENT) physician to ensure suitability for the hyperbaric chamber.

Exclusion Criteria:

* chronic obstructive pulmonary disease, malignancy
* cardiac pacemakers, or any disorder that lead to ulcers other than diabetes
* chronic peripheral arterial disease.

Ages: 55 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2025-06-01 (Actual); Primary Completion 2025-07-15 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Ulcer volume using Saline injection method | 4 weeks

SECONDARY OUTCOMES:
Tcpo2 at ulcer edge using Pulse Oximeter | 4 weeks
Emg pre and at end (Sensory NCS (Sural nerve) | 4 weeks

CONTACTS AND LOCATIONS:
Locations (1):
- Modern University For Technology and Information, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided